CLINICAL TRIAL: NCT01988246
Title: Prevention of Macular Edema In Patients With Diabetic Retinopathy Undergoing Cataract Surgery
Acronym: PROMISE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rishi Singh (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Rishi Singh, staff surgeon / Sponsor-Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PROMISE Trial
Record Dates: First submitted 2013-10-30; First posted 2013-11-20 (Estimated); Results first posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetes; Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus | interventions — aflibercept; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham Injection (Sham Comparator): Patients will be sequentially randomized to treatment with a "sham" injection at the time of surgery. The sham injection is accomplished by pressing an empty syringe against the eye wall without penetration. This will be administered post cataract excision by the Prinicipal Investigator. The patient will be masked as to which Arm they are assigned.
  Interventions: Drug: Sham
- Intravitreal Aflibercept Injection (Active Comparator): Patients will be sequentially randomized to treatment with Aflibercept 2 mg via intravitreal injection (0.05 mL or 50 microliters) at the time of surgery. This will be administered post cataract excision by the Principal Investigator. The patient will be masked as to which Arm they are assigned.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Patients will be assigned to treatment with 2 mg intravitreal Aflibercept injection (0.05 mL or 50 microliters) administered at the time of surgery (post cataract excision) or sham injection.
  Other Names: Eylea
  Arms: Intravitreal Aflibercept Injection
Drug: Sham — Sham injection. No actual injection. No medication is used.
  Arms: Sham Injection

SUMMARY:
To determine the safety and efficacy of intravitreal Aflibercept (Eylea) injection in patients with diabetic retinopathy in the prevention of macular edema following cataract surgery.

DETAILED DESCRIPTION:
Diabetic retinopathy patients who are at risk of developing macular edema (defined as ≥ 30 % increase from pre-operative baseline in central subfield macular thickness) within 90 days following cataract surgery. Diabetic patients are defined as those who have either Type 1 or Type 2 diabetes. The patients must have either mild, moderate, or severe non proliferative retinopathy or treated proliferative retinopathy. Patients must be 18 years of age and older, of any race and either sex, requiring cataract extraction with planned implantation of a posterior chamber intraocular lens into the lens capsule.

ELIGIBILITY:
Inclusion Criteria:

* A patient must meet the following criteria to be eligible for inclusion in the study:

  1. Must be 18 years of age and older, of any race and either sex, who have a cataract, and are planning to undergo cataract extraction by phacoemulsification with the implantation of a posterior chamber intraocular lens into the lens capsule
  2. History of Type I or Type II diabetes
  3. NPDR: non-proliferative diabetic retinopathy (mild, moderate, or severe) or inactive proliferative disease in the study eye as defined by the International Clinical Diabetic Retinopathy Disease Severity Scale
  4. Willing and able to comply with clinic visits and study-related procedures
  5. Patients must be able to understand and sign an informed consent that has been approved by an Institutional Review Board (IRB)
  6. Central subfield macular thickness ≤ 320 μm in the study eye prior to cataract surgery as determined by SD-OCT and confirmed by the reading center
  7. Absence of clinically significant macular edema (CSME) in the study eye as detected by clinical exam
  8. Patients must have visual acuity of 20/20-20/200

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from the study:

1. Signs of vitreomacular traction or epiretinal membrane in the study eye as detected by reading center or investigator
2. Current or previous ocular disease in the study eye that in the opinion of the investigator may confound assessment of the macula, the retina, or central vision other that diabetic retinopathy
3. Active proliferative diabetic retinopathy in the study eye
4. Planned multiple procedures for study eye during the cataract/IOL implantation surgery (e.g., trabeculectomy, corneal transplant)
5. Patients who have received corneal transplants in the study eye
6. Patients with current or history of chronic or recurrent ocular infections or inflammation in the study eye
7. Patients with a visually nonfunctional fellow eye based upon the assessment by the investigator
8. Patients who are immunocompromised (e.g., patients receiving chemotherapy irradiation therapy, patients with AIDS, leukemia, or cachexia) or patients receiving dialysis
9. Use of medications known to affect the macula, including hydroxychloroquinine (Plaquenil) and phenothiozines (e.g., thioridazine [Mellaril], chloropromazine [Thorazine]) or supplemental niacin ≥3 grams/day
10. Use of systemic steroids, NSAIDS (non-steroidal anti-inflammatory drugs), anti-VEGF agents within 7 days prior to surgery (through study exit). Daily doses of aspirin, up to 325 mg, will be permitted.
11. Use of topical ocular NSAIDS and steroids, in the study eye, within 7 days prior to surgery
12. Treatment with intraocular or periocular steroids in the study eye within 3 months prior to surgery
13. Focal photocoagulation for the treatment of diabetic macular edema in the study eye within 6 months of the pre-operative baseline visit (Note: peripheral retina treatment for retinal tear or lattice degeneration is permitted)
14. Intravitreal anti-VEGF (vascular endothelial growth factor) treatment in the study eye within 6 months of the pre-operative baseline visit
15. Patients with a known hypersensitivity to NSAIDs or steroids or any component of the study medication.
16. Use of a topical ophthalmic prostaglandin (e.g., TRAVATAN, XALATAN) within 4 days of surgery through study exit
17. Any concurrent intraocular condition in the study eye that, in the opinion of the investigator, could require either medical or surgical intervention during the 90 day study period.
18. Any concurrent ocular condition in the study eye which, in the opinion of the investigator, could either increase the risk to the patient beyond what is to be expected from standard procedures of intraocular injection, or which otherwise may interfere with the injection procedure or with evaluation of efficacy or safety.
19. Pregnant or breast-feeding women -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12; Primary Completion 2018-04-25 (Actual); Study Completion 2020-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rishi Singh, M.D., Principal Investigator — Cole Eye Institute, Cleveland Clinic
Locations (1):
- Cole Eye Institute, Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham Injection | Intravitreal Aflibercept Injection
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Injection | Intravitreal Aflibercept Injection | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Customized [Mean (Full Range); unit: years] | 66 [47 to 80] | 66 [53 to 80] | 66 [47 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 5 | 9 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 6 | 10 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Ocular and Non-Ocular Adverse Events
Description: Number of participants with ocular and non-ocular adverse events (AEs) in both treatment arms.
Time Frame: Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Injection | Intravitreal Aflibercept Injection
Number analyzed (Participants) | 15 | 15
Participants
  At least 1 Ocular Adverse Event | 11 | 10
  At least 1 Non-Ocular Adverse Event | 5 | 3

2. Secondary Outcome: Change From Baseline in Best-Corrected Visual Acuity (BCVA) Score
Description: Change from baseline in best-corrected visual acuity (BCVA) score and BCVA score at Day 90 as measured by ETDRS (early treatment diabetic retinopathy study) There were no sub scales used. These are common methods for ophthalmology studies to report their findings. The scale provided is the Electronic-Early Treatment in Diabetic Retinopathy Scale (E-ETDRS) best corrected visual acuity scale. Values that are higher are considered better and values that are lower are considered worse. Minimum E-ETDRS was 24 E-ETDRS letters and maximum E-ETDRS was 80 E-ETDRS letters.
Time Frame: Day 90
Measure: Mean (95% Confidence Interval); unit: Number of Letters Read Correctly
Arm/Group | Sham Injection | Intravitreal Aflibercept Injection
Number analyzed (Participants) | 15 | 15
Number of Letters Read Correctly | 8.52 [4.26 to 12.78] | 9.88 [5.54 to 14.22]

3. Other Pre Specified Outcome: Change From Baseline in Retinal Thickness
Description: The change in macular edema as measured by SD-OCT (spectral domain ocular coherence tomography)at 90 days
Time Frame: Day 90
Measure: Mean (95% Confidence Interval); unit: Microns
Arm/Group | Sham Injection | Intravitreal Aflibercept Injection
Number analyzed (Participants) | 15 | 15
Microns | 50.32 [14.49 to 86.15] | 18.48 [0.87 to 36.09]

ADVERSE EVENTS:
Time Frame: Up to 90 days following each surgery
Arm/Group | Sham Injection | Intravitreal Aflibercept Injection
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15 | 3/15
Other Adverse Events (participants affected / at risk) | 14/15 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Injection (N=15) | Intravitreal Aflibercept Injection (N=15)
Paracentesis (Eye disorders) | 0 | 2
Cough/Vomiting (Gastrointestinal disorders) | 0 | 1
Rash and Swelling on Limbs (Skin and subcutaneous tissue disorders) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Injection (N=15) | Intravitreal Aflibercept Injection (N=15)
Foreign Body Sensation (Eye disorders) | 3 | 3 — Foreign Body Sensation of Eye
Corneal Edema (Eye disorders) | 0 | 1 — Corneal Swelling
Eye Irritation/Pain (Eye disorders) | 2 | 2 — Eye irritation and pain
Eye Itching (Eye disorders) | 1 | 2 — Eye Itching
Lacrimation Increased (Eye disorders) | 1 | 1 — Eye Tearing
Blurred Vision (Eye disorders) | 4 | 2 — Blurred Vision
Photophobia (Eye disorders) | 3 | 0 — Light Sensitivity
Floaters (Eye disorders) | 4 | 2 — Floaters in Vision

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT01988246/Prot_SAP_000.pdf
  • Informed Consent Form (2015-05-08): https://cdn.clinicaltrials.gov/large-docs/46/NCT01988246/ICF_001.pdf